CLINICAL TRIAL: NCT02810041
Title: Randomized Controlled Double-blind Clinical Trial for the Effect of Yoghurts Enriched in XXS vs Without XXS on the Evolution of Weight in Overweight Subjects Aged 50 to 65 Years.
Brief Title: Effect of Yoghurts Enriched With XXS (Mixture of Natural Polyphenolic Compounds and Plant Extracts) on the Evolution of Weight in Overweight Subjects
Acronym: VITALIM Senior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: VAN WYMELBEKE SENOBLE 2013
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- yoghurts enriched with XXS (Experimental)
  Interventions: Dietary Supplement: yoghurts enriched with XXS
- yoghurts non enriched with XXS (Placebo Comparator)
  Interventions: Dietary Supplement: yoghurts non enriched with XXS

INTERVENTIONS:
Dietary Supplement: yoghurts enriched with XXS
  Arms: yoghurts enriched with XXS
Dietary Supplement: yoghurts non enriched with XXS
  Arms: yoghurts non enriched with XXS

SUMMARY:
Overweight and obesity are public health problems worldwide. Even though heredity may be one of the causes the diseases, the vast majority of cases is rather linked to a sedentary lifestyle associated or not with a low-variety, high-calorie diet. Many diets and slimming methods propose low-calorie meals or physical exercise, and the consequences of these are sometimes negative with advancing age (muscle wasting). Certain studies have shown the efficacy of foods with antioxidant properties on the reduction of blood pressure, Low Density Lipoprotein (LDL)-cholesterol and weight or on the distribution of fat mass-lean mass. The investigators put forward the hypothesis that the daily consumption of two yoghurts containing XXS, a mixture of natural polyphenolic compounds -rich in quercetin- from plant extracts, could lead to weight loss, a better fat mass-lean mass distribution and an improvement in markers of oxidative stress in overweight persons aged 50 to 65 years.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged between 50 and 65 years;
* who have provided written consent;
* and are covered by national health insurance;
* with a stable weight for 6 months and no intention to begin a diet in the coming three months;
* with a Body Mass Index (BMI) between 25 and 29.9 kg/m2 and a waist circumference > 80 cm in women and > 94cm in men (thresholds of the International Diabetes Federation, IDF);
* who consume dairy products such as yoghurts;
* and do not have more than two of the following risk factors of metabolic syndrome: known history of hypertension (>130/85mmHg), hypocholesterolemia High Density Lipoprotein HDL (< 0.4 g/L men and 0.5 g/L women), hypertriglyceridemia (>1.5 g/L), diabetes (> 1.1 g/L);
* presenting C Reactive Protein (CRP) < 6mg/L.

Exclusion Criteria:

* adults under guardianship
* persons following a prescribed of self-prescribed diet;
* whose behaviour may interfere with the consumption of the active dairy product (more than 4h of physical activity a week, smoking more than 10 cigarettes a day, more than 2 glasses of alcohol a day, Consuming more than one bar of dark chocolate a day, 10 cups of coffee/day, 5 large cups of tea/day, supplementation with vitamins (A, C, E…), oligoelements or minerals (Se, Zn, Ca…), enriched dairy products or any supplements containing Dietary Foods for Specialized Medical Purposes (ADFMS) .

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2015-05-27 (Actual); Study Completion 2015-05-27 (Actual)

PRIMARY OUTCOMES:
Bodyweight | Change from baseline bodyweight at day 60, day100 at 105 in the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Champmaillot Geriatric Department, Dijon, France